CLINICAL TRIAL: NCT00204503
Title: An Open Label Pilot Study Evaluating Safety and Efficacy of Divalproex Sodium (Depakote ER) in Patients With Bipolar I or II Depression and Alcohol Abuse or Dependence.
Brief Title: Open-Label Depakote ER in Patients With Bipolar I or II Depression and Alcohol Abuse or Dependence
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 03-048; FRS 467640
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2015-03-31 (Estimated); Status verified 2015-03

CONDITIONS: Bipolar I or II Depression and Alcohol Abuse or Dependence
Keywords: Bipolar I or II; Depression; Alcohol Abuse or Dependence; Mental Health Issues
MeSH Terms: conditions — Alcoholism; Depression | interventions — Valproic Acid

INTERVENTIONS:
Drug: Depakote ER

SUMMARY:
The purpose of this study is to determine if Divalproex Sodium can be used to Treat and Prevent Depression in Patients with Bipolar Disorder who have Comorbid Alcohol Dependence/Abuse.

DETAILED DESCRIPTION:
Over half of all patients with bipolar disorder have comorbid substance abuse. The most common substance of abuse is alcohol, which is most commonly associated with the depressed phase of the illness. Although there are available treatments for bipolar depression, no studies have been done to evaluate efficacy in bipolar patients with comorbid substance abuse disorders. Given the independent open-label evidence for efficacy and safety of divalproex sodium in alcohol abuse and bipolar depression, divalproex sodium is the most likely candidate for potential success in bipolar depressed patients with comorbid alcohol abuse or dependence. The purpose of this study is to determine if Divalproex Sodium can be used to Treat and Prevent Depression in Patients with Bipolar Disorder who have Comorbid Alcohol Dependence/Abuse.

ELIGIBILITY:
Inclusion Criteria:

* MADRS >= 20 at screen and 18 at baseline
* YMRS =< 11 at screen and baseline
* DMS-IV criteria for past manic or hypomanic episode based on the SCID
* DSM-VI criteria for alcohol dependence or abuse based on the SCID.
* Alcohol dependence/abuse confirmed by corroboration from family member
* Negative urine pregnancy test

Exclusion Criteria:

* Inability to give informed consent
* Inability to give reliable assessment of alcohol consumption
* Evidence of alcohol consumption one week prior to baseline
* Liver function tests greater than 3X upper limit of normal at screen
* History of active hepatitis or hepatic encephalopathy
* History of pancreatitis
* History of adverse reaction to divalproex sodium
* History of seizure other than directly associated w/prior alcohol withdrawl
* History of major head trauma with LOC > 10 min. or skull fracture
* Hisotry of hypertension or neurologic illness
* If female, not practicing an effective form of birth control

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2003-06; Study Completion 2005-05

PRIMARY OUTCOMES:
Primary Efficacy Measures for this study are: Percent change in MADRS from baseline score to study endpoint; Percent of days heavy drinking from 120 days prescreen to study end point; and Percent of subjects successfully completing outpatient detox.

SECONDARY OUTCOMES:
Secondary Efficacy Measures for this study are: Percent change in IDS-SR and YMRS from baseline to end of week 16.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Stone, M.D., Principal Investigator — The University of Texas Medical Branch, Galveston
Locations (1):
- University of Texas Medical Branch, Galveston, Texas, United States